CLINICAL TRIAL: NCT05060900
Title: Hand Ligament Reconstructions With Knee Collateral Ligament Allografts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Kulber, MD, Director of Hand and Upper Extremity Surgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000044
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hand Injuries; Wrist Injuries; Ligament Injury; Ligament Rupture; Ligament Avulsion
Keywords: hand ligament injury, wrist ligament injury
MeSH Terms: conditions — Hand Injuries; Wrist Injuries; Fractures, Avulsion

STUDY DESIGN:
Intervention Model Description: All patients enrolled in the study will undergoing their ligament reconstruction procedure with allograft ligament.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand and Wrist Ligament Reconstruction with Allograft Ligament (Experimental): Participants will undergo surgery for hand and wrist ligament reconstruction using allograft ligament.
  Interventions: Procedure: Ligament Reconstruction with Allograft Ligament

INTERVENTIONS:
Procedure: Ligament Reconstruction with Allograft Ligament — Patients will undergo surgery for hand and wrist ligament reconstruction using allograft ligament.

SUMMARY:
The purpose of this study is to review the clinical outcomes following hand ligament reconstruction surgery using allograft (cadaveric) knee collateral ligaments. Currently, there is no standard procedure or devices used for hand ligament reconstruction surgery, although most techniques use some form of autograft (patients' own tissue) for the reconstruction. We believe that the use of allograft ligaments in reconstruction may eliminate the pain associated with procuring the patients' own tissue for the procedure, and prove to be a viable and preferred alternative to the multiple techniques currently used.

The main procedures of this study include wrist and hand ligament reconstruction surgery (for wrist scapholunate (SL) ligaments, thumb ulnar collateral ligaments (UCL), and finger proximal interphalangeal (PIP) joint collateral ligaments) using allograft ligament, and subsequent follow up appointments where measurements and questionnaires will be completed to evaluate how hand function is doing after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Have symptomatic injuries to either their finger PIP collateral ligaments, thumb UCL ligaments, or wrist SL ligaments and have failed non-operative management for the above ligament injuries (thus eligible for operative reconstruction)
* Age over 18 years

Exclusion Criteria:

* Presence of any other current injury in that limb
* Presence of advanced arthrosis in that limb
* Presence of fixed joint deformity in that limb
* Presence of instability in that limb due to bony or articular instability
* Presence of instability in that limb due to inflammatory arthrosis
* Is under 18 years of age
* Lacks the capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in functional outcome, as measured by the quick Disabilities of the Arm, Shoulder and Hand (qDASH) questionnaire | Baseline, post-surgery 6 week, post-surgery 6 month, post-surgery 1 year
  The qDASH questionnaire asks about symptoms of upper extremity disability as well as the ability to perform certain activities. It generates a score from 0 to 100, with higher scores indicating greater severity of disability.
Change from baseline in pain, as measured by the Visual Analog Scale (VAS) | Baseline, post-surgery 6 week, post-surgery 6 month, post-surgery 1 year
  The VAS generates a scale from 0 to 100 with 0 indicating no pain and higher scores indicating greater pain.
Change from baseline in key pinch strength, as measured with a pinch gauge. | Baseline, post-surgery 6 week, post-surgery 6 month, post-surgery 1 year
  A pinch gauge is a device that measures key pinch strength in units of pounds or Newtons.
Change from baseline in grip strength, as measured with a Jamar hand dynamometer. | Baseline, post-surgery 6 week, post-surgery 6 month, post-surgery 1 year
  A Jamar hand dynamometer is a device that measures grip strength in units of pounds or Newtons.
Change from baseline in wrist and finger range of motion angles. | Baseline, post-surgery 6 week, post-surgery 6 month, post-surgery 1 year
  Range of motion to be assessed includes wrist extension, wrist flexion, wrist ulnar deviation, wrist radial deviation, finger proximal interphalangeal joint flexion and extension, thumb metacarpophalangeal joint flexion and extension, thumb abduction and adduction.
Change from baseline in wrist and finger radiographs. | Baseline, post-surgery 6 week, post-surgery 6 month, post-surgery 1 year
  Radiographic images obtained can help indicate the success of surgery by demonstrating joint stability.

CONTACTS AND LOCATIONS:
Overall Officials: David Kulber, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No